CLINICAL TRIAL: NCT07368829
Title: Feasibility and Safety of Artificial Intelligence-Driven Autonomous Registration in Robotic Navigational Bronchoscopy
Brief Title: AI-Driven Autonomous Registration in Robotic Bronchoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Director, Department of Thoracic Surgery, Ruijin Hospital, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: RTS-030
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lung Nodules; Bronchoscopy; Localization Efficiency
Keywords: Artificial Intelligence; Robotic Bronchoscopy; Pulmonary Nodule

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autonomous registration group (Experimental): All participants in this arm will undergo robotic navigational bronchoscopy and pulmonary nodule localization performed using the Langhe Bronchoscopy Robot System. The key intervention is the use of artificial intelligence (AI)-driven autonomous registration technology to automatically align the pre-operative chest CT images with the real-time bronchoscopic anatomy prior to the procedure. This process aims to reduce reliance on the conventional, operator-dependent manual registration. Physicians will supervise the entire process and perform necessary manual intervention if the AI registration is unsatisfactory or for safety reasons.
  Interventions: Device: AI-driven autonomous registration

INTERVENTIONS:
Device: AI-driven autonomous registration — All participants in this arm will undergo robotic navigational bronchoscopy and pulmonary nodule localization performed using the Langhe Bronchoscopy Robot System. The key intervention is the use of artificial intelligence (AI)-driven autonomous registration technology to automatically align the pre-operative chest CT images with the real-time bronchoscopic anatomy prior to the procedure. This process aims to reduce reliance on the conventional, operator-dependent manual registration. Physicians will supervise the entire process and perform necessary manual intervention if the AI registration is unsatisfactory or for safety reasons.

SUMMARY:
This study aims to evaluate the feasibility and safety of an artificial intelligence (AI)-driven autonomous registration technology in robotic navigational bronchoscopy. A total of 20 patients with pulmonary nodules requiring localization will be enrolled. The Langhe Bronchoscopy Robot System equipped with AI-based autonomous registration software will be used. Primary outcomes include the success rate of autonomous registration and the rate of manual intervention during the process. Secondary outcomes encompass registration time, complication rates, and nodule localization success.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Radiologically confirmed pulmonary nodules requiring preoperative localization.
* Scheduled for robotic navigational bronchoscopy using the Bronchoscopy Robot System.
* Willing to provide written informed consent.

Exclusion Criteria:

* Severe cardiopulmonary dysfunction (e.g., FEV1 < 30% predicted).
* Coagulopathy or anticoagulation therapy that cannot be safely interrupted.
* Pregnancy or lactation.
* Inability to tolerate bronchoscopy under general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Autonomous registration success rate | Intraoperative
  Proportion of registrations completed independently by the AI algorithm without manual intervention.
Manual intervention rate during autonomous registration | Intraoperative
  The proportion of cases requiring manual adjustment by the physician during the registration process.

SECONDARY OUTCOMES:
Time consumed for autonomous registration | Intraoperative
Complication rate during autonomous registration | Immediate post-procedure to 24 hours
  Complication rate during autonomous registration (e.g., bleeding, pneumothorax)
Localization success rate of pulmonary nodules | Intraoperative
  The proportion of successful bronchoscope arrivals at the target nodule after registration.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No